CLINICAL TRIAL: NCT00474006
Title: A RANDOMIZED COMPARISON OF TWO DIFFERENT DOSAGES OF DAUNORUBICIN IN INDUCTION TREATMENT OF ACUTE MYELOGENOUS LEUKEMIA
Brief Title: High Dose Daunorubicin Vs. Standard Dose Daunorubicin in Induction Treatment of AML
Acronym: ADcomparison
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cooperative Study Group A for Hematology (Network)
Responsible Party: COSAH, Cooperative Study Group A for Hematology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C-006
Record Dates: First submitted 2007-05-15; First posted 2007-05-16 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-06

CONDITIONS: ACUTE MYELOGENOUS LEUKEMIA
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Daunorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- arm I (Active Comparator): Cytarabine 200 mg/m2/d civ x 7 days Daunorubicin 45 mg/m2/d civ x 3 days
  Interventions: Drug: arm II

INTERVENTIONS:
Drug: arm II — Cytarabine 200 mg/m2/d civ x 7 days Daunorubicin 90 mg/m2/d civ x 3 days
  Other Names: regular dose of Daunorubicin (Arm I); higher dose of Daunorubicin (ArmI)

SUMMARY:
Determine the effects of escalated dose of daunorubicin in induction treatment of adult patients with acute myelogenous leukemia who are younger than 60 years of age.

DETAILED DESCRIPTION:
1. Induction chemotherapy

   * For patients randomized to receive regular dose of Daunorubicin (Arm I) will be given Cytarabine 200 mg/m2/day by continuous iv infusion over 24 hours daily for 7 days along with Daunorubicin 45 mg/m2/day by continuous iv infusion over 24 hours daily for 3 days.
   * For patients randomized to receive higher dose of Daunorubicin (Arm II) will be given Cytarabine 200 mg/m2/day by continuous iv infusion over 24 hours daily for 7 days along with Daunorubicin 90 mg/m2/day by continuous iv infusion over 24 hours daily for 3 days.
2. Reinduction chemotherapy

   * Bone marrow aspiration and biopsy will be performed on day 14 of induction chemotherapy. If the bone marrow is hypoplastic and contains no more than 5% blast cells, further chemotherapy will be deferred and the marrow examination will be repeated at the time of ANC ≥ 1,500/μl and platelets ≥ 100,000/μl in the peripheral blood for the evaluation of complete remission. If more than 5% blast cells persist or if the marrow cellularity in the biopsy specimen exceeds 15%, a course of reinduction chemotherapy will be given.
   * Reinduction chemotherapy consists of Cytarabine 200 mg/m2/day by continuous iv infusion over 24 hours daily for 5 days along with Daunorubicin 45 mg/m2/day by continuous iv infusion over 24 hours daily for 2 days in both arms.
3. Postremission therapy

   * The same postremission therapy will be given to the patients in both arms.
   * Four courses of Cytarabine 3 g/m2 will be administered in a 3-hour iv infusion every 12 hours (twice daily) on days 1, 3, and 5 for a total of six doses per course. After the four courses of Cytarabine therapy, patients will receive two monthly treatments with Cytarabine (200 mg/m2/day by a 3-hour iv infusion for 5 days) and Daunorubicin (45 mg/m2 by rapid iv infusion on the first treatment day).
   * If patients have HLA-matched sibling or unrelated donors, allogeneic stem cell transplantation will be performed.
   * A complete remission will be defined as ≤ 5% blasts in a normocellular bone marrow with ANC ≥ 1,500/μl and platelets ≥ 100,000/μl in the peripheral blood and the disappearance of all blasts in bone marrow.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed AML or RAEB
* 15 years of age or older, but younger than 60 years of age
* Adequate hepatic and renal function
* Normal cardiac function with LVEF ≥ 50% on MUGA scan or echocardiogram
* Written informed consent

Exclusion Criteria:

* promyelocytic leukemia or chronic myelogenous leukemia
* significant infection
* prior chemotherapy history for leukemia

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 398 (Actual)
Dates: Start 2001-08; Primary Completion 2008-08 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Toxicities, complete remission rate, duration of complete remission, disease-free survival, overall survival | 10years
  The effects will be evaluated in terms of toxicities, complete remission rate, duration of complete remission, disease-free survival, and overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Je Hwan Lee, professor, Principal Investigator — Asan Medical Center, ROK
Locations (1):
- Asan Medical Center, Seoul, Songpa-gu, South Korea

REFERENCES:
- [Derived] Lee JH, Joo YD, Kim H, Bae SH, Kim MK, Zang DY, Lee JL, Lee GW, Lee JH, Park JH, Kim DY, Lee WS, Ryoo HM, Hyun MS, Kim HJ, Min YJ, Jang YE, Lee KH; Cooperative Study Group A for Hematology. A randomized trial comparing standard versus high-dose daunorubicin induction in patients with acute myeloid leukemia. Blood. 2011 Oct 6;118(14):3832-41. doi: 10.1182/blood-2011-06-361410. Epub 2011 Aug 9. PMID 21828126